CLINICAL TRIAL: NCT01531309
Title: An Open-Label, Parallel-Group Study to Compare the Pharmacokinetics, Safety and Tolerability of a Single Sublingual 1 mg Dose of AGO178 in Subjects With Mild and Moderate Hepatic Impairment With That in Matched Healthy Control Subjects
Brief Title: Pharmacokinetics of AGO178 in Participants With Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAGO178C2102
Record Dates: First submitted 2012-02-03; First posted 2012-02-10 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Impairment
Keywords: Liver impairment; Major Depression Disorder; Sublingual tablet
MeSH Terms: interventions — agomelatine

ARMS (3):
- Mild Hepatic Impaired Participants (Experimental): Mild hepatic impaired participants will receive a single sublingual dose of AGO178, 1 milligram (mg) on Day 1.
  Interventions: Drug: AGO178
- Moderate Hepatic Impaired Participants (Experimental): Moderate hepatic impaired participants will receive a single sublingual dose of AGO178, 1 mg on Day 1.
  Interventions: Drug: AGO178
- Healthy Participants Matched by Aged, Gender and Body Mass Index (BMI) (Experimental): Healthy participants matched by aged, gender and BMI will receive a single sublingual dose of AGO178, 1 mg on Day 1.
  Interventions: Drug: AGO178

INTERVENTIONS:
Drug: AGO178 — AGO178 is administered as a sublingual tablet.
  Other Names: Agomelatine

SUMMARY:
AGO178 was developed for the treatment of depression. A new formulation is being tested in the present study: a tablet to be placed and dissolved under the tongue (sublingual tablet). The goal of this trial was to study the pharmacokinetics of agomelatine given as sublingual tablet in participants with liver impairment and to compare the results to those of healthy volunteers who receive the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with liver disease confirmed within 3 months of screening.
* If liver impairment is caused by alcohol use, participants must have abstained from alcohol use within 3 months of study start.
* Participants must satisfy criteria for Child- Pugh Class A or B.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless using effective contraception during the study.
* Donation or loss of 400 millilitres (mL) or more of blood within eight (8) weeks prior to initial dosing.
* Significant illness within the two weeks prior to the dosing.
* Participants with Child-Pugh alterations due to a non-liver disease (e.g. cancer or treatment related weight loss).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2011-09-02 (Actual); Study Completion 2011-09-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of AGO178 | Predose, 2 minute (min) , 5 min , 10 min, 20 min, 30 min, 45 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 12h, 24h, 36h Post dose
  Blood samples will be collected at various time points on day 1 and day 2
Area Under the Plasma Curve (AUC) of AGO178 | Predose, 2 min , 5 min , 10 min, 20 min, 30 min, 45 min, 1h, 1.5h, 2h, 3h, 4h, 6h, 12h, 24h, 36h Post dose
  Blood samples will be collected at various time points on day 1 and day 2

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Baseline and Day 8
  Adverse events will be based on evaluation of physical signs, electrocardiograms and clinical laboratory assessments (clinical chemistry, hematology, urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States